CLINICAL TRIAL: NCT06831175
Title: Phase II Study of PD-1 Inhibitor Combined With Apatinib and Mitotane in the Treatment of Advanced Adrenal Cortical Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1549
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Adrenal Cortical Carcinoma; Adrenal Cortical Cancer; Adrenal Cancer
Keywords: Camrelizumab; Mitotane; Apatinib; Advanced Adrenal Cortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Gland Neoplasms | interventions — camrelizumab; apatinib; Mitotane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Camrelizumab in combination with apatinib and mitotane (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Apatinib; Drug: mitotane

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab was administered 200mg IV every 3 weeks.
Drug: Apatinib — Apatinib was administered 250 mg PO QD.
  Other Names: Rivoceranib; YN968D1
Drug: mitotane — Mitotane is administered orally and plasma concentration was measured. The target steady-state plasma concentration is 14-20 mg/L.

SUMMARY:
Adrenocortical carcinoma (ACC) is a rare aggressive malignant tumor. According to the literature, the 5-year survival rate of ACC is 12%-47%. For patients with advanced ACC, mitotane alone or combined with traditional chemotherapy was the first-line standard treatment, but its progression-free survival was only about 1 year. The efficacy of mitotane monotherapy is approximately 10% to 30%. FIRM-ACT trial reported an objective response rate (ORR) of 23.2% for etoposide, doxorubicin, cisplatin, and mitotane (EDP-M) chemotherapy regimen. Our phase II study found that PD-1 inhibitor camrelizumab and apatinib showed impressive clinical data in the second-line treatment of relapsed and metastatic ACC patients. The aim of this study is to evaluate the efficacy and safety of PD-1 inhibitor camrelizumab combined with apatinib and mitotane in advanced ACC, and to explore a new treatment strategy for patients with advanced ACC.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological diagnosis of adrenocortical carcinoma;
2. Patients with unresectable advanced adrenocortical carcinoma who have not received first-line standard treatment;
3. Age ≥18 years old, ≤70 years old;
4. No gender limit;
5. Eastern Cooperative Oncology Group (ECOG) score 0-1;
6. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1);
7. Major organ function within 28 days before treatment, meeting the following criteria:

   - Blood routine test criteria (without blood transfusion within 14 days) : Hemoglobin (HB) ≥80g/L Absolute neutrophil count (ANC) ≥1.5×10^9/L Platelet (PLT) ≥80×10^9/L

   - Biochemical tests must meet the following criteria: Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN or ≤5 ULN if liver metastases are present Serum creatinine (Cr) ≤1.5 ULN or creatinine clearance (CCr)≥60 ml/min

   - Coagulation testing requires the following criteria: International normalized ratio (INR) or prothrombin time (PT) ≤1.5 ULN Activated partial thromboplastin time (APTT) ≤1.5 ULN (if the patient is anticoagulated, as long as the PT and APTT are within the intended therapeutic range)

   - Cardiac markers and natriuretic peptide (BNP) ≤ULN;
8. Women of childbearing age should agree that they must use a contraceptive method (such as an intrauterine device, contraceptive pill, or condom) during the study and for 120 days after the study; Patients had a negative serum or urine pregnancy test within 7 days before study entry and had to be non-lactating; Men should consent to patients who must use contraception during the study and for 6 months after the end of the study period;
9. Study participants provided written informed consent and were willing and able to follow planned visits, study treatments, laboratory tests, and other experimental procedures.

Exclusion Criteria:

1. A history of other malignant tumors within the past 5 years or at the same time, except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and thyroid papillary carcinoma;
2. Known allergic reactions to other monoclonal antibodies, active ingredient of mitotane, active ingredient of apatinib and or any excipients;
3. CNS metastases with clinical symptoms such as brain edema, requiring hormonal intervention, or progression of brain metastases;
4. Patients who received potent CYP3A4 inhibitor treatment within one week before enrollment or a potent CYP3A4 inducer treatment within two weeks before the first use of study drug;
5. Patients with hypertension not well controlled by antihypertensive drug therapy alone (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
6. NYHA class III-IV congestive heart failure;
7. Occurrence of arterial/venous thrombosis events within 1 year before enrollment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), myocardial infarction, unstable angina pectoris, deep vein thrombosis, and pulmonary embolism;
8. QT interval > 500 ms;
9. Prior systemic immunosuppressive therapy;
10. Prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies;
11. TKI treatment within 2 weeks before the first dose;
12. Participating in other interventional drug clinical trials within 4 weeks before the first dose;
13. Received an antineoplastic vaccine or a live vaccine within 4 weeks before the first dose of study drug;
14. Major surgery or major trauma within 4 weeks before the first dose of study medication;
15. Had a serious infection (CTCAE > 2) within 4 weeks before the first dose of study drug, such as severe pneumonia requiring hospitalization, bacteremia, and infectious complications; The presence of active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first dose of the study drug, or the need for treatment with oral or intravenous antibiotics (excluding prophylactic antibiotics) on baseline chest imaging.
16. Have an active autoimmune disease, a history of autoimmune disease (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes); Autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type 1 diabetes on stable doses of insulin; However, patients with vitiligo or childhood asthma/allergies that had been cured and did not need any intervention in adulthood were excluded.
17. Have a history of immunodeficiency, including being HIV positive or having other acquired or congenital immunodeficiency disorders, or having a history of organ or bone marrow transplantation;
18. A history of non-infectious pneumonia;
19. Active pulmonary tuberculosis infection detected by medical history or CT examination, or a history of active pulmonary tuberculosis infection within 1 year before enrollment or patients who had a history of active pulmonary tuberculosis infection 1 year ago but had not received formal treatment;
20. Subjects with active hepatitis (HBV DNA≥2000 IU/ml or 10000 copies/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA above the detection limit of the assay);
21. A known history of psychotropic drug abuse, alcohol abuse, and drug use;
22. Have GI bleeding symptoms and risk of bleeding;
23. Are pregnant or lactating;
24. Have medical history, disease, treatment, or laboratory abnormalities that may interfere with the results of the trial or prevent the subject from participating fully in the study, or the investigator believes that participation in the study is not in the subject's best interest.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | up to 24 months
  The rate of complete response and partial response.

SECONDARY OUTCOMES:
disease-free survival | up to 60 months
  The time from the administration of the first dose to first disease progression or death.
progression-free survival | up to 60 months
  The time from the commencement of therapy to the first evidence of disease progression or death.
incidence of adverse events | up to 60 months
  Graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu YC, Wei ZG, Wang JJ, Pei YY, Jin J, Li D, Li ZH, Liu ZR, Min Y, Li RD, Yang L, Liu JY, Wei Q, Peng XC. Camrelizumab plus apatinib for previously treated advanced adrenocortical carcinoma: a single-arm phase 2 trial. Nat Commun. 2024 Nov 29;15(1):10371. doi: 10.1038/s41467-024-54661-9. PMID 39609453
- [Background] Habra MA, Stephen B, Campbell M, Hess K, Tapia C, Xu M, Rodon Ahnert J, Jimenez C, Lee JE, Perrier ND, Boraddus RR, Pant S, Subbiah V, Hong DS, Zarifa A, Fu S, Karp DD, Meric-Bernstam F, Naing A. Phase II clinical trial of pembrolizumab efficacy and safety in advanced adrenocortical carcinoma. J Immunother Cancer. 2019 Sep 18;7(1):253. doi: 10.1186/s40425-019-0722-x. PMID 31533818
- [Background] Raj N, Zheng Y, Kelly V, Katz SS, Chou J, Do RKG, Capanu M, Zamarin D, Saltz LB, Ariyan CE, Untch BR, O'Reilly EM, Gopalan A, Berger MF, Olino K, Segal NH, Reidy-Lagunes DL. PD-1 Blockade in Advanced Adrenocortical Carcinoma. J Clin Oncol. 2020 Jan 1;38(1):71-80. doi: 10.1200/JCO.19.01586. Epub 2019 Oct 23. PMID 31644329
- [Background] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- [Background] Berruti A, Terzolo M, Sperone P, Pia A, Della Casa S, Gross DJ, Carnaghi C, Casali P, Porpiglia F, Mantero F, Reimondo G, Angeli A, Dogliotti L. Etoposide, doxorubicin and cisplatin plus mitotane in the treatment of advanced adrenocortical carcinoma: a large prospective phase II trial. Endocr Relat Cancer. 2005 Sep;12(3):657-66. doi: 10.1677/erc.1.01025. PMID 16172198
- [Background] Tang Y, Liu Z, Zou Z, Liang J, Lu Y, Zhu Y. Benefits of Adjuvant Mitotane after Resection of Adrenocortical Carcinoma: A Systematic Review and Meta-Analysis. Biomed Res Int. 2018 Jun 4;2018:9362108. doi: 10.1155/2018/9362108. eCollection 2018. PMID 29967789
- [Background] Abiven G, Coste J, Groussin L, Anract P, Tissier F, Legmann P, Dousset B, Bertagna X, Bertherat J. Clinical and biological features in the prognosis of adrenocortical cancer: poor outcome of cortisol-secreting tumors in a series of 202 consecutive patients. J Clin Endocrinol Metab. 2006 Jul;91(7):2650-5. doi: 10.1210/jc.2005-2730. Epub 2006 May 2. PMID 16670169
- [Background] Icard P, Goudet P, Charpenay C, Andreassian B, Carnaille B, Chapuis Y, Cougard P, Henry JF, Proye C. Adrenocortical carcinomas: surgical trends and results of a 253-patient series from the French Association of Endocrine Surgeons study group. World J Surg. 2001 Jul;25(7):891-7. doi: 10.1007/s00268-001-0047-y. PMID 11572030
- [Background] Else T, Kim AC, Sabolch A, Raymond VM, Kandathil A, Caoili EM, Jolly S, Miller BS, Giordano TJ, Hammer GD. Adrenocortical carcinoma. Endocr Rev. 2014 Apr;35(2):282-326. doi: 10.1210/er.2013-1029. Epub 2013 Dec 20. PMID 24423978
- [Background] Allolio B, Fassnacht M. Clinical review: Adrenocortical carcinoma: clinical update. J Clin Endocrinol Metab. 2006 Jun;91(6):2027-37. doi: 10.1210/jc.2005-2639. Epub 2006 Mar 21. PMID 16551738